CLINICAL TRIAL: NCT02299635
Title: PHASE 2 STUDY OF SINGLE-AGENT PF-03084014 IN PATIENTS WITH ADVANCED TRIPLE-NEGATIVE BREAST CANCER WITH OR WITHOUT GENOMIC ALTERATIONS IN NOTCH RECEPTORS
Brief Title: A Study Evaluating PF-03084014 In Patients With Advanced Breast Cancer With Or Without Notch Alterations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on June 24th, 2015 due to change in strategy of PF-03084014 development. There were no safety/efficacy concerns behind the decision.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A8641020; 2014-002286-30 (EudraCT Number)
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Triple Negative Breast Neoplasms
Keywords: PF-03084014; Notch Alterations
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — nirogacestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-03084014 (Experimental): PF-03084014 will be administered orally, continuously, twice daily at 150 mg, but the dose can be reduced to 100 mg or 80 mg.
  Interventions: Drug: PF-03084014

INTERVENTIONS:
Drug: PF-03084014 — Tablet, 10 mg, twice a day.
Drug: PF-03084014 — Tablet, 50 mg, twice a day
Drug: PF-03084014 — Tablet, 100 mg, twice a day

SUMMARY:
This study is designed to evaluate the preliminary anti-tumor activity and tolerability of PF-03084014 when administered as a single agent in the treatment of patients with advanced triple receptor-negative breast cancer (mTNBC) harboring genomic alterations in Notch receptors (NA+), and in a smaller subset of mTNBC patients whose tumor tests negative for genomic alterations in Notch receptors (NA-)

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of triple negative breast cancer (TNBC) with evidence of a) metastatic or b) locally recurrent advanced disease that is not amenable to resection or radiotherapy with curative intent.
* Availability of an original diagnostic tumor tissue or the most recent metastatic tumor biopsies (archival biopsy or de novo biopsy) and a peripheral blood sample for Notch receptors genomic profiling

Exclusion Criteria:

* Known brain metastases.
* Prior treatment with gamma secretase inhibitor or other Notch signaling inhibitor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2016-01-14 (Actual); Study Completion 2016-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (18):
  - Stanford Cancer Institute, Stanford, California
  - Stanford Hospital and Clinics, Stanford, California
  - Stanford Women's Cancer Center, Stanford, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Brigham and Women's Hospital (BWH), Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Medical Group, Paramus, New Jersey
  - Valley Medical Group, Westwood, New Jersey
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center Sleepy Hollow, Sleepy Hollow, New York
- Debreceni Egyetem, Klinikai Kozpont, Onkologiai Intezet, Debrecen, Hungary
- Italy (2):
  - Presidio Ospedaliero Vito Fazzi, Lecce
  - Istitutio Europeo di Oncologia, Milan
- Poland (3):
  - Vesalius, Krakow
  - Vesalius Poradnia Onkologiczna i Hematologiczna, Krakow
  - Szpital Kliniczny Przemienienia Panskiego, Uniwersutetu Medycznego im. Karola Marcinkowskiego, Poznan
- Spain (9):
  - Complejo Hospitalario Universitario A Coruna (Hospital Teresa Herrera), A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Instituto Catalan de Oncologia de L'Hospitalet de Llobregat (ICO), Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Ross Hall Hospital, Glasgow, Scotland
  - The Royal Marsden NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8641020&StudyName=A%20Study%20Evaluating%20PF-03084014%20In%20Patients%20With%20Advanced%20Breast%0ACancer%20With%20Or%20Without%20Notch%20Alterations

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-03084014: PF-03084014 at the starting dose of 150 mg twice daily (BID) (in the form of one 100-mg and one 50-mg tablet) was administered orally BID continuously in 21-day cycles until disease progression, patient refusal of further treatment, or unacceptable toxicity, whichever occurred first.
Period: Overall Study
Arm/Group | PF-03084014
Started | 19
Completed | 0
Not Completed | 19
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Global deterioration of health status | 1
Not completed — Objective progression or relapse | 10
Not completed — Withdrawal by Subject | 2
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | PF-03084014
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (OR) Rate in Participants With Advanced Triple Receptor-Negative Breast Cancer (mTNBC) Harboring Activating Genomic Alterations in Notch Receptors (NA+)
Description: OR status based on assessment of confirmed complete remission (CR) or confirmed partial remission (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1). CR: Complete disappearance of all target lesions with the exception of nodal disease and all target nodes decreased to normal size (short axis less than [<]10 millimeter [mm]). PR: Greater than or equal to (>=)30% decrease under baseline of the sum of diameters of all target measurable lesions. OR=CR+PR.
Time Frame: Cycle 3 Day 1, Cycle 5 Day 1, and every 6 weeks for subsequent cycles ntil disease progression, patient refusal for further follow up, or start of another anti-cancer treatment, whichever occurred first.
Population: Data for this outcome measure was not collected due to early termination of this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

2. Secondary Outcome: OR Rate in Participants With mTNBC Whose Tumors Tested Negative for Eenomic Alterations in Notch Receptor (NA-)
Description: OR status based on assessment of confirmed CR or confirmed PR according to RECIST 1.1. CR: Complete disappearance of all target lesions with the exception of nodal disease and all target nodes decreased to normal size (short axis <10 mm). PR: >=30% decrease under baseline of the sum of diameters of all target measurable lesions. OR=CR+PR.
Time Frame: as for outcome 1
Population: Data for this outcome measure was not collected due to early termination of this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-Free Survival (PFS) in Participants With NA+ or NA mTNBC
Description: The period from study entry until disease progression, death, whichever occurred first as per RECIST version 1.1.
Time Frame: 2 years
Population: Data for this outcome measure was not collected due to early termination of this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response (DR) in Participants With NA+ or NA mTNBC
Description: Time from the first documentation of objective tumor response to objective tumor progression or death due to any cause. DR was calculated for the subgroup of patients with a confirmed objective tumor response. Objective Progression (PD): 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy), with a minimum absolute increase of 5 mm.
Time Frame: 2 years
Population: Data for this outcome measure was not collected due to early termination of this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

5. Secondary Outcome: One-Year Survival Probability in Participants With NA+ or NA mTNBC
Description: Overall survival (OS) status (alive or not) at 1 year after study entry. The the survival probability at 1 year was summarized as a product limit estimator based on the Kaplan-Meier method to account for censored events.
Time Frame: 1 year
Population: Data for this outcome measure was not collected due to early termination of this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival (OS) in Participants With NA+ or NA mTNBC
Description: OS was the duration from enrollment to death. For participants who are alive, overall survival was censored at the last contact.
Time Frame: 2 years
Population: Data for this outcome measure was not collected due to early termination of this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

7. Secondary Outcome: Type of Notch Genomic Alterations in Participants With NA+ mTNBC
Description: Type of notch genomic alterations identified by NGS assay in patients with NA+ mTNBC
Time Frame: 2 years
Population: Data for this outcome measure was not collected due to early termination of this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

8. Secondary Outcome: Pre-dose Serum Concentration (Ctrough) for PF-03084014
Time Frame: Day 1 of Cycle 1, 2, 3, and 5
Population: Due to study termination, no PK analyses were performed for this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

9. Secondary Outcome: Pharmacodynamic (PD) Effects of PF-03084014 in Tumor Specimens and Peripheral Blood
Description: Original diagnostic tumor tissue or the most recent metastatic tumor (archival or de novo biopsy), plasma, and peripheral blood samples were collected for biomarker assessments of circulating analytes, immunohistochemistry for notch receptors expression, expression of notch pathway components and modulators, mutational analysis of pathway and disease associated genes.
Time Frame: Day 1 of Cycle 1, 2, 3, and 5
Population: Due to study termination, no PD analyses were performed for this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

10. Secondary Outcome: Alterations in Genes, Proteins, and RNAs Relevant to the Notch Signaling Pathway, to TNBC Biology, and to Sensitivity/Resistance to PF-03084014 in Tumor Specimens and Peripheral Blood.
Description: as for outcome 9
Time Frame: Day 1 of Cycle 1, 2, 3, and 5
Population: Due to study termination, no PD analyses were performed for this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were defined as all deaths, regardless of cause, from treatment start until 28 days after the last dose and non-fatal events occurring after treatment start regardless of cause, up until 28 days after the last dose or until start of new anti-cancer treatment, whichever was first.
Time Frame: 2 years
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014
Number analyzed (Participants) | 19
participants
  Number of Participants with AEs | 18
  Number of Participants with SAEs | 6

12. Secondary Outcome: Number of Participants With Treatment-Emergent AEs by CTCAE Grade
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. AEs were defined according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 2 years
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014
Number analyzed (Participants) | 19
participants
  Any AEs, Grade 1 | 1
  Any AEs, Grade 2 | 5
  Any AEs, Grade 3 | 9
  Any AEs, Grade 4 | 1
  Any AEs, Grade 5 | 2

13. Secondary Outcome: Number of Participants With Laboratory Test (Hematology) Abnormalities
Description: Number of participants with CTCAE version 4.03 grade 1 to 4 hematological test abnormalities.
Time Frame: Day 1 of Cycles 1, 2, 3, 4, 5, and subsequent cycles.
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014
Number analyzed (Participants) | 19
participants
  Anemia | 12
  Lymphocyte count increased | 0
  Lymphopenia | 11
  Neutrophils (absolute) | 0
  Platelets | 3
  White blood cells | 4

14. Secondary Outcome: Number of Participants With Laboratory Test (Chemistry) Abnormalities
Description: Number of participants with CTCAE version 4.03 grade 1 to 4 chemistry test abnormalities
Time Frame: Day 1 and Day 15 of Cycles 1, 2, 3, 4, 5, and subsequent cycles up to Cycle 8 and Day 8 of Cycle 1
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014
Number analyzed (Participants) | 19
participants
  Alanine aminotransferase | 5
  Alkaline phosphatase | 6
  Aspartate aminotransferase | 9
  Bilirubin (total) | 1
  Creatine kinase | 1
  Creatinine | 13
  Gamma glutamyl transferase | 1
  Hypercalcemia | 3
  Hyperglycemia | 13
  Hyperkalemia | 3
  Hypermagnesemia | 1
  Hypernatremia | 0
  Hypoalbuminemia | 8
  Hypocalcemia | 4
  Hypoglycemia | 1
  Hypokalemia | 5
  Hypomagnesemia | 3
  Hyponatremia | 6
  Hypophosphatemia | 14

15. Secondary Outcome: Number of Participants With Laboratory Test (Urinalysis) Abnormalities
Description: Number of participants with CTCAE version 4.03 grade 1 to 4 urinalysis test abnormalities for urine protein.
Time Frame: Day 1 of Cycle 1
Population: The safety analysis set included all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-03084014
Number analyzed (Participants) | 19
participants | 2

16. Secondary Outcome: Number of Notch Genomic Alterations in Participants With NA+ mTNBC
Description: Number of notch genomic alterations identified by NGS assay in patients with NA+ mTNBC
Time Frame: 2 years
Population: Data for this outcome measure was not collected due to early termination of this study.
Arm/Group | PF-03084014
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | PF-03084014
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03084014 (N=19)
Disease progression (General disorders) | 1
Pyrexia (General disorders) | 1
Lung infection (Infections and infestations) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusional state (Psychiatric disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03084014 (N=19)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Eye discharge (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Oral pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 1
Chest pain (General disorders) | 2
Fatigue (General disorders) | 8
Mucosal inflammation (General disorders) | 3
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 5
Conjunctivitis (Infections and infestations) | 3
Gastroenteritis viral (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 1
Blood chloride decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Carbon dioxide increased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Protein total increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 7
Hypouricaemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tumour exudation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Rash macular (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated prematurely based on project re-prioritization by the Sponsor and was not due to any safety concerns or regulatory actions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.